CLINICAL TRIAL: NCT00797108
Title: A Phase 2 Randomized, Double-blind, Double-dummy Efficacy, Safety And Tolerability Study Of Iv Sulopenem With Switch To Oral Pf-03709270 Compared To Ceftriaxone With Step Down To Amoxicillin/Clavulanate Potassium (Augmentin) In Subjects With Community Acquired Pneumonia (Cap) Requiring Hospitalization
Brief Title: A Study Of Intravenous Sulopenem And Oral PF-03709270 In Community Acquired Pneumonia That Requires Hospitalization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8811020; 2008-006307-23 (EudraCT Number)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — sulopenem; Ceftriaxone; Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Loading dose of IV sulopenem with switch to oral PF-03709270
  Interventions: Drug: sulopenem and PF-03709270
- 2 (Experimental): IV sulopenem with switch to oral PF-03709270
  Interventions: Drug: Sulopenem and PF-03709270
- 3 (Active Comparator): IV ceftriaxone with switch to oral amoxicillin/clavulanate potassium comparator
  Interventions: Drug: Ceftriaxone and amoxicillin/clavulanate

INTERVENTIONS:
Drug: sulopenem and PF-03709270 — Sulopenem - 600 mg infused over 1 hour, single loading dose and switch to oral PF-03709270 - 1000 mg twice a day
  Arms: 1
Drug: Sulopenem and PF-03709270 — Sulopenem - 600 mg infused over 1 hour twice daily for a minimum of 2 days and switch to oral PF-03709270 - 1000 mg twice a day
  Arms: 2
Drug: Ceftriaxone and amoxicillin/clavulanate — IV ceftriaxone (2g) infused over 30 minutes QD (once daily) for minimum of 2 days Step down oral amoxicillin/clavulanate potassium suspension (400 mg/5 ml) BID (every 12 hours)
  Arms: 3

SUMMARY:
The purpose of this study is to test if intravenous sulopenem and an oral drug, PF-03709270 are safe and effective in patients that are hospitalized with community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female patients 18 years of age or older.
* Female patients of childbearing potential must not be pregnant.
* Must exhibit at least two pre-specified clinical symptoms/signs of pneumonia.
* Must require hospitalization for the pneumonia.
* Chest Xray must be suggestive of a pneumonia.

Exclusion Criteria:

* Hospital or ventilator associated pneumonia.
* Patients with cystic fibrosis, pneumocystis carinii pneumonia or active tuberculosis.
* Previous treatment for the current pneumonia episode received for more than 24 hours.
* Allergies to penems or beta lactams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (10):
  - eStudySite, Inc., Chula Vista, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - eStudySite, Inc., Oceanside, California
  - Tri-City Medical Center, Oceanside, California
  - Medical Arts Associates, Ltd, Moline, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Infectious Disease Minneapolis Limited, Minneapolis, Minnesota
  - Summa Health System, Akron, Ohio
  - Utah Valley Pulmonary Clinic, Provo, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
- Infection Management Services, Building 17, Level 1, Brisbane, Queensland, Australia
- Canada (3):
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - Hamilton Health Sciences- McMaster Site, Hamilton, Ontario
  - Hamilton Health Sciences - Henderson Site, Hamilton, Ontario
- Poland (7):
  - Oddzial Chorob Wewnetrznych i Gastroenterologii, Bialystok
  - Oddzial Chorob Pluc, Brzesko
  - Kliniczny Oddzial Gruzlicy i Chorob Pluc, Krakow
  - Oddzial Kliniczny Pulmonologii i Alergologii, Lodz
  - Oddzial Pulmonologiczny III, Poznan
  - Oddzial Pulmonologiczny, Proszowice
  - II Oddzial Chorob Wewnetrznych, Warsaw
- Asan Medical Center, Division of Infectious Diseases, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8811020&StudyName=A%20Study%20Of%20Intravenous%20Sulopenem%20And%20Oral%20PF-03709270%20In%20Community%20Acquired%20Pneumonia%20That%20Requires%20Hospitalization

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulopenem (Single Intravenous Dose) and PF-03709270: Single loading dose of sulopenem 600 milligram (mg) intravenous infusion over 1 hour, followed by oral PF-03709270 (5*200 mg tablets) 12 hours after loading dose, twice daily during in-patient period (minimum of 2 days equivalent on intravenous dose or as per investigator's discretion), along with placebo intravenous infusion over 1 hour and then twice daily for minimum of 3 doses, followed by placebo intravenous infusion over 30 minutes once daily for minimum of 2 doses. After in-patient period, switched to oral PF-03709270 1000 mg (5*200 mg tablets) twice daily along with oral placebo suspension twice daily. Total treatment duration of 7 to 10 days was at the discretion of the investigator.
- Sulopenem (Multi Intravenous Dose) and PF-03709270: Sulopenem 600 mg intravenous infusion over 1 hour twice daily for minimum of 4 doses, followed by oral placebo tablets 12 hours after first intravenous dose, twice daily during in-patient period (minimum of 2 days equivalent on intravenous dose or as per investigator's discretion) along with placebo intravenous infusion over 30 minutes once daily for minimum of 2 doses. After in-patient period, switched to oral PF-03709270 1000 mg (5*200 mg tablets) twice daily along with oral placebo suspension twice daily. Total treatment duration of 7 to 10 days was at the discretion of the investigator.
- Ceftriaxone and Amoxicillin/Clavulanate: Ceftriaxone 2 gram (g) intravenous infusion over 30 minutes once daily for minimum of 2 doses, followed by oral placebo tablets 12 hours after first intravenous dose, twice daily during in-patient period (minimum of 2 days equivalent on intravenous dose or as per investigator's discretion) along with placebo intravenous infusion over 1 hour twice daily for minimum of 4 doses. After in-patient period, stepped down to oral amoxicillin/clavulanate potassium suspension (800 mg/10 milliliter) twice daily along with oral placebo tablets twice daily. Total treatment duration of 7 to 10 days was at the discretion of the investigator.
Period: Overall Study
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Started | 12 | 11 | 12
Treated | 10 | 11 | 12
Completed | 8 | 9 | 6
Not Completed | 4 | 2 | 6
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Did Not Meet Entrance Criteria | 0 | 1 | 0
Not completed — Global Deterioration of Health Status | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Other | 0 | 0 | 2
Not completed — Randomized but not Treated | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who received at least 1 dose of double blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate | Total
Number analyzed (Participants) | 10 | 11 | 12 | 33
Age, Customized [Number; unit: participants]
  18 to 44 years | 0 | 1 | 0 | 1
  45 to 64 years | 2 | 4 | 5 | 11
  greater than or equal to (>=) 65 years | 8 | 6 | 7 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 15
  Male | 4 | 5 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response at Test of Cure (TOC) Visit
Description: Clinical response (CR) was based primarily on global assessment of clinical presentation of participant made by investigator at evaluation time point. At TOC (7 to 14 days after end of treatment [EOT]) CR was evaluated as "cure"=resolution of clinical signs and symptoms related to the acute infection, or clinical improvement in which no additional antibiotics were deemed necessary when compared to baseline; "failure"=persistence or progression of baseline signs and symptoms of pneumonia (for example: body temperature, white blood cell [WBC] count, respiratory rate, auscultatory findings, cough, sputum production), development of new pulmonary or extrapulmonary clinical findings consistent with active infection and those participants that were not assessed for clinical response due to early discontinuation; "indeterminate"=extenuating circumstances precluded classification to 1 of the above.
Time Frame: 7 to 14 days after end of treatment
Population: Clinically evaluable: all ITT participants who received at least 80% of study drug, no concomitant systemic antibiotic with activity against relevant pathogens, diagnosed with pneumonia as defined by protocol inclusion criteria, assignment of pneumonia severity index (PSI) score III (low: score range 71-90)-IV(high: score range 91-130).
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 8 | 8
percentage of participants
  Cure | 90.0 | 87.5 | 62.5
  Failure | 10.0 | 12.5 | 25.0
  Indeterminate | 0 | 0 | 12.5
Statistical Analysis 1: Comparison: Sulopenem (Single Intravenous Dose) and PF-03709270 vs Ceftriaxone and Amoxicillin/Clavulanate; Two-sided 80% confidence interval (CI) for the difference in the clinical cure response rates between treatement group and the comparator was formed using the exact methods; Test type: Superiority or Other; Clinical Cure Difference = 27.5, 80% CI 2-sided [-4.0 to 55.3]
Statistical Analysis 2: Comparison: Sulopenem (Multi Intravenous Dose) and PF-03709270 vs Ceftriaxone and Amoxicillin/Clavulanate; Two-sided 80% CI for the difference in the clinical cure response rates between treatement group and the comparator was formed using the exact methods; Test type: Superiority or Other; Clinical Cure Difference = 25.0, 80% CI 2-sided [-13.1 to 57.9]

2. Secondary Outcome: Percentage of Participants With Clinical Response at End of Treatment (EOT) and Follow-up Visit
Description: CR was based primarily on global assessment of clinical presentation of participant made by investigator at evaluation time point. At EOT (Day 7 to 10) and follow-up (15 to 28 days after EOT), CR was evaluated as "cure"=resolution of clinical signs and symptoms related to the acute infection, or clinical improvement in which no additional antibiotics were deemed necessary when compared to baseline; "failure"=persistence or progression of baseline signs and symptoms of pneumonia, development of new pulmonary or extrapulmonary clinical findings consistent with active infection and those participants that were not assessed for clinical response due to early discontinuation; with additional CR evaluated as "improvement"= of few not all signs and symptoms of pneumonia when compared to baseline and no additional antibacterial treatment required at EOT and "indeterminate"=extenuating circumstances precluded classification to 1 of the above at follow-up.
Time Frame: EOT (Day 7 to 10) , Follow-up (15 to 28 days after EOT)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 8 | 8
percentage of participants
  EOT: Cure | 60.0 | 75.0 | 75.0
  EOT: Improvement | 30.0 | 25.0 | 12.5
  EOT: Failure | 10.0 | 0.0 | 12.5
  Follow-up: Cure | 90.0 | 87.5 | 62.5
  Follow-up: Failure | 0.0 | 0.0 | 12.5
  Follow-up: Indeterminate | 10.0 | 12.5 | 25.0

3. Secondary Outcome: Number of Participants With Microbiological Response at Test of Cure (TOC) Visit
Description: Microbiological response assessed at participant level. Eradication=the absence of the original pathogens from the post-treatment TOC culture of specimen from the original site of infection. Presumed eradication=the complete resolution of signs and symptoms associated with cessation of culturable specimen (for example, sputum). Persistence=the presence of the original pathogen in the post-treatment TOC culture specimen from the original site of infection. Presumed persistence=in a participant who was judged to be a clinical failure and a culture of specimen was not possible or was not done, it was presumed that there was persistence of the pathogen. Not applicable microbiologic response included participants that did not have post-treatment microbiologic cultures due to early discontinuation. Data reported for eradication is combination of eradication and presumed eradication data and data reported for persistence is combination of persistence and presumed persistence data.
Time Frame: 7 to 14 days after EOT
Population: Microbiologic clinically evaluable population included all microbiologic ITT participants (all ITT participants in whom a pathogen was isolated at baseline) who also met criteria for the clinically evaluable subset.
Measure: Number; unit: participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 4 | 5 | 4
participants
  Eradication | 4 | 4 | 3
  Persistence | 0 | 0 | 0
  Not Applicable | 0 | 1 | 1

4. Secondary Outcome: Change From Baseline in Community Acquired Pneumonia (CAP) Symptom Questionnaire at Test of Cure (TOC) and Follow-up Visit
Description: The CAP Symptom Questionnaire was a participant reported questionnaire administered by interview. It consisted of 12 items (coughing, chest pains, shortness of breath, sweating, chills, headache, nausea, muscle pain, lack of appetite, trouble concentrating, trouble sleeping, and fatigue). Depending on if the participant had or not had symptoms/problems, they were asked how much they had been bothered by the symptoms/problems over the previous 24 hours. CAP items were rated on the 6-point response scale (0 = participant did not have symptom/problem: 1 = not at all, 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely; if the participant had the symptom/problem and were bothered). All 12 items score were summed and averaged to produce a CAP symptom score (range, 0 to 6). High values indicated poorer outcomes (higher symptom bothersomeness).
Time Frame: Baseline, TOC (7 to 14 days after end of treatment), Follow-up (15 to 28 days after EOT)
Population: Clinically evaluable population. Here 'n' signifies participants evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 8 | 8
units on a scale
  Baseline (n=10, 8, 8) | 2.17 (0.70) | 2.75 (1.01) | 2.57 (0.65)
  Change at TOC (n=9, 7, 6) | -1.43 (0.85) | -2.02 (1.23) | -1.74 (0.86)
  Change at Follow-up Visit (n=10, 8, 8) | -1.39 (0.86) | -1.89 (1.08) | -1.52 (1.00)

5. Other Pre Specified Outcome: Number of Participants Who Died
Time Frame: Baseline up to 15 to 28 days after EOT
Population: ITT population included all randomized participants who received at least 1 dose of double blind study drug.
Measure: Number; unit: participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 11 | 12
participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Test Findings
Description: Criteria for laboratory abnormalities: hemoglobin (Hb), hematocrit, red blood cell (RBC) (less than [<] 0.8*lower limit of normal [LLN]); reticulocyte (absolute and percentage) (<0.5*LLN or greater than [>] 1.5*upper LN [ULN]); platelet (<0.5*LLN or >1.75*ULN); white blood cell (WBC) (<0.6*LLN or >1.5*ULN); lymphocyte, neutrophil (<0.8*LLN or >1.2*ULN); eosinophil, monocyte, basophil (>1.2*ULN); bilirubin (BR) (>1.5*ULN); aspartate and alanine aminotransferase, gamma-glutamyl transpeptidase, alkaline phosphatase, lactate dehydrogenase (>3.0*ULN); total protein, albumin (<0.8*LLN or >1.2*ULN);blood urea nitrogen, creatinine (>1.3*ULN); sodium (<0.95*LLN or >1.05*ULN); potassium, chloride, calcium, magnesium, bicarbonate (<0.9*LLN or >1.1*ULN); glucose (<0.6*LLN or >1.5*ULN); urine (pH [<4.5 or >8], glucose, protein, blood, ketone [>=1]). Total number of participants with abnormal laboratory values were reported.
Time Frame: Baseline up to 15 to 28 days after EOT
Population: ITT population included all randomized participants who received at least 1 dose of double blind study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 11 | 11
participants | 7 | 8 | 9

7. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: A physical examination included an examination of the general appearance, skin, heart, head, eyes, ears, nose, throat, breasts, abdomen, musculoskeletal, neck, neurological, extremities, and others. Criteria for abnormal physical findings were based on investigator's discretion.
Time Frame: Last observation (up to 15-28 days after EOT, approximately 38 days)
Population: ITT population included all randomized participants who received at least 1 dose of double blind study drug.
Measure: Number; unit: participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 10 | 11 | 12
participants | 0 | 1 | 0

8. Other Pre Specified Outcome: Number of Participants With Categorical Change From Baseline in Vital Signs
Description: Participants who met the categorical criteria for increase in vital signs data were reported. Categorical criteria for increase from baseline vital signs data: supine and sitting systolic blood pressure (BP) of greater than or equal to (>=) 30 millimeter of mercury (mmHg); supine and sitting diastolic BP of >=20 mmHg.
Time Frame: Baseline up to 15 to 28 days after EOT
Population: ITT population included all randomized participants who received at least 1 dose of double blind study drug. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies participants evaluable for this measure for specified category for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 7 | 6 | 6
participants
  Supine Systolic BP >=30 mmHg (n=3, 5, 4) | 0 | 2 | 1
  Sitting Systolic BP >=30 mmHg (n=7, 6, 6) | 2 | 1 | 1
  Supine Diastolic BP >=20 mmHg (n=3, 5, 4) | 0 | 2 | 2
  Sitting Diastolic BP >=20 mmHg (n=7, 6, 6) | 4 | 1 | 0

9. Other Pre Specified Outcome: Population Pharmacokinetics
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study.
Time Frame: 0.5 to 1 hours, 1.5 to 3 hours, 3 to 5 hours after initiation of first intravenous dose; 0.5 to 2.5 hours, 4 to 6 hours following administration of oral dose on the day of IV to oral switch (minimum of 2 days equivalent on intravenous dose)
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)

10. Other Pre Specified Outcome: Number of Participants With Healthcare Resource Utilization
Description: Healthcare resource utilization was to be evaluated using the assessment of the following: date and duration of index admission, duration of hospitalization, date of discharge, location of discharge, type/length of treatment inside and outside of the hospital, healthcare professional visits outside of the hospital, emergency room visits, and other hospitalizations.
Time Frame: Baseline up to 15 to 28 days after EOT
Population: This assessment was not performed due to the small sample size and hence data for this outcome measure is not reported.
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sulopenem (Single Intravenous Dose) and PF-03709270 | Sulopenem (Multi Intravenous Dose) and PF-03709270 | Ceftriaxone and Amoxicillin/Clavulanate
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/11 | 2/12
Other Adverse Events (participants affected / at risk) | 6/10 | 6/11 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulopenem (Single Intravenous Dose) and PF-03709270 (N=10) | Sulopenem (Multi Intravenous Dose) and PF-03709270 (N=11) | Ceftriaxone and Amoxicillin/Clavulanate (N=12)
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyothorax (Infections and infestations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulopenem (Single Intravenous Dose) and PF-03709270 (N=10) | Sulopenem (Multi Intravenous Dose) and PF-03709270 (N=11) | Ceftriaxone and Amoxicillin/Clavulanate (N=12)
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Application site erythema (General disorders) | 1 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.